CLINICAL TRIAL: NCT06396000
Title: Prolonged Stay in the Pediatric PACU
Brief Title: Factors Analysis Related to Prolonged Stay in the Pediatric Post-Anesthesia Care Unit(PACU)
Acronym: PACU
Status: Not yet recruiting | Type: Observational
Sponsor: Saiqiang Guo (Other)
Responsible Party: Sponsor-Investigator, Saiqiang Guo, Senior nurse, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: FARPSPP
Record Dates: First submitted 2024-04-23; First posted 2024-05-02 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia; Adverse Effect
Keywords: Post-anesthesia care unit; Risk factors; Pediatrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine which factors contribute to prolonged stay of children in the PACU.

DETAILED DESCRIPTION:
Studying the factors associated with prolonged stay of children in the PACU is of great significance to the medical team, as it can improve the quality and speed of anesthesia recovery, not only in line with the concept of accelerated rehabilitation surgery, but also through intervention and optimization of specific factors to improve the efficiency of children's postoperative discharge from the PACU, reduce the incidence of complications, lower medical costs, and increase patient and family satisfaction. Therefore, this study aims to explore the factors associated with prolonged stay of children in the PACU through retrospective analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-18 years old; Child entering the Pediatric Post-Anesthesia Care.
* Emergency surgery; Pediatric patients with incomplete medical history; Pediatric patients requiring postoperative ICU care; Pediatric patients with preoperative altered consciousness; Neurological disorders; Severe liver, kidney, lung, and heart diseases.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patient entering the Pediatric Post-Anesthesia Care.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Anesthesia Plan Selection | Day 1
  Anesthesia options include general anesthesia, combined anesthesia, pure intravenous anesthesia, and nerve block anesthesia.
Pain Score | Day 1
  Evaluate pain using the Visual Analog Scale (VAS): 0 points: no pain; 1-3 points: mild pain; 4-6 points: moderate pain; 7-10 points: severe pain.
Complications in PACU | Day 1
  Nausea, vomiting, chills, pain, agitation
American Society of Anesthesiologists（ASA） | Day 1
  ASA I: Patients in good health, without systemic disease. ASA II: Patients with mild systemic disease, not significantly limiting daily activity.
  ASA III: Patients with severe systemic disease, with definite functional limitation.
  ASA IV: Patients with severe systemic disease that is a constant threat to life.
  ASA V: Moribund patients who are not expected to survive without the operation. ASA VI: Brain-dead patients whose organs are being removed for donation.
The medication usage in PACU | Day 1
  Morphine, Propofol, Ketorolac, Fentanyl

SECONDARY OUTCOMES:
The use of PCA（Patient-Controlled Analgesia）in PACU | Day 1
  PCA usage statistics，yes or no